CLINICAL TRIAL: NCT06600126
Title: Supporting Evidence-based Responses to Emotional Needs in Emphysema
Acronym: SERENE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Henry Ford Health System (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 852619; R01NR020819 (NIH)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: COPD
Keywords: Pulmonary Disease; Coping Skills; Psychological Distress; Mixed Methods
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coping Skills Training (Experimental)
  Interventions: Behavioral: Coping Skills Training
- COPD Education (Experimental)
  Interventions: Behavioral: COPD Education

INTERVENTIONS:
Behavioral: Coping Skills Training — The Coping Skills Training arm will consist of 12 weekly 30-minute sessions via videoconferencing or phone. A trained research staff member will deliver sessions that focus on building coping skills for patients with COPD, such as progressive relaxation training, pleasant activity scheduling, and building communication skills. Caregivers will also participate, learning how to support the patient in using these skills. Participants will complete assignments between sessions to reinforce their learning. Additionally, participants will receive a Coping Skills Training workbook.
  Arms: Coping Skills Training
Behavioral: COPD Education — The COPD Education arm will consist of 12 weekly 10-minute sessions via videoconferencing or phone. A trained research staff member will provide scripted general support and encouragement without using specific psychoeducational techniques. Caregivers will also participate. Additionally, participants will receive a COPD Education workbook with material from The COPD Foundation, which is also available on the Foundation's website. This program augments usual care, providing an attention control for comparison.
  Arms: COPD Education

SUMMARY:
The goal of this clinical trial is to understand how a Coping Skills Training program can reduce depression and anxiety in people with chronic obstructive pulmonary disease (COPD), particularly those who face health disparities, including those with low income, different racial backgrounds, or those living in rural areas. The main questions it aims to answer are:

* How does the Coping Skills Training program help reduce stress and anxiety in patients?
* What causes variations in the effectiveness of the Coping Skills Training program?
* What are the barriers and facilitators to the uptake of the Coping Skills Training program?

Researchers will compare a 12-week Coping Skills Training program with a COPD Education program to see if the training leads to better health outcomes for participants.

Participants will:

* Take part in weekly 30-minute sessions for 12 weeks if assigned to the Coping Skills Training group.
* Take part in weekly 10-minute sessions for 12 weeks if assigned to the COPD Education group.
* Complete surveys before, during, and after the intervention.
* Patients and caregivers, including those who chose not to enroll, as well as clinicians, will be invited to participate in interviews to share their perspectives.

DETAILED DESCRIPTION:
Social environments, including family structure and function, shape patients' care and outcomes. Yet the role of family caregivers in chronic illness care is often unrecognized or undervalued even when critically relevant. For example, psychological distress is highly prevalent among patients with chronic obstructive pulmonary disease (COPD). COPD affects more than 212 million people worldwide, annual US medical costs are over $49 billion, and groups experiencing health disparities are most affected. Family caregivers, patients, and clinicians identify emotional symptoms and coping as critical priorities in COPD care. Psychological distress is strongly associated with poor quality of life and clinical outcomes for patients with COPD, such as more frequent exacerbations and higher post-discharge mortality. Yet affected patients rarely receive psychological care, particularly patients who face barriers to behavioral health care access. Integrating families into approaches to reduce patients' psychological distress is likely to improve outcomes and equity.

The investigators' overarching objective is to reduce the burden of chronic illness on patients and families. The central hypothesis is that improving patients' coping skills and caregivers' ability to coach patients in use of these skills will improve patients' outcomes. The existing evidence amongst patients with COPD is strongest for non- pharmacological interventions for psychological distress, but fails to represent diverse study populations. High-quality family relationships (i.e., cohesion, problem solving, and communication) are associated with better clinical outcomes. Among patients with COPD, better family relationship quality is associated with reduced psychological distress and improved self-management and dyspnea. Coping Skills Training is a scalable intervention that uses cognitive-behavioral skills to teach patient-caregiver dyads how to respond to the many emotional, physical, functional, and psychosocial consequences of COPD. In an NIH-funded trial of 326 dyads, Coping Skills Training improved patients' psychological and health-related quality of life more than an educational control. Yet, the mechanisms of the intervention's success remain unknown and the prior work underrepresented groups experiencing health disparities. Filling these critical knowledge gaps is an urgent need that will allow the investigators to refine and scale effective and efficient interventions addressing this critical need.

The investigators propose a randomized clinical trial to test putative treatment mechanisms through which the Coping Skills Training program administered to patients with COPD and their family caregivers improves outcomes. Outpatients with COPD who screen positive for psychological distress will be randomized in a 2:1 ratio to participate in a 12-week program with a caregiver, either a Coping Skills Training program (i.e., weekly 30-minute protocolized sessions delivered by a behavioral health specialist) or COPD Education program (i.e., weekly 10-minute sessions without coping skills).

ELIGIBILITY:
Inclusion Criteria:

Patients

* Be at least 18 years of age
* Have a documented diagnosis of COPD and confirmation of obstructive lung disease by spirometry (American Thoracic Society/European Respiratory Society guidelines) or radiology (imaging report indicating emphysematous changes)
* Score greater than or equal to 8 during baseline screening using the PHQ-8
* Identify an adult caregiver to participate with them
* Have the ability to access a telephone or videoconferencing call up to once weekly (for approximately 30 minutes) for 12 sessions of the study intervention
* Spoken proficiency in Spanish and/or English

Caregivers

* Be at least 18 years of age
* Have the ability to access a telephone or videoconferencing call up to once weekly (for approximately 30 minutes) for 12 weeks

Exclusion Criteria:

Patients

* Has significant dementia or cognitive impairment
* Documentation in the EHR that the COPD diagnosis has not yet been disclosed to the patient
* Is under the ongoing care of a licensed behavioral health clinician
* Requires immediate referral to specialized behavioral health management

Caregivers

* Has significant dementia or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-03-05 (Estimated)

PRIMARY OUTCOMES:
Patient Psychological Distress | Baseline, 14 weeks
  Patient psychological distress will be measured using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 consists of 9 items, with total scores ranging from 0 to 27. Higher scores indicate greater distress.

SECONDARY OUTCOMES:
Patient Psychological Distress (Secondary Outcome) | Baseline, 7 weeks, 26 weeks
  Patient psychological distress will be measured as a secondary outcome using the Patient Health Questionnaire-9 (PHQ-9) after 7 weeks and 14 weeks. As described above, the PHQ-9 consists of 9 items, with total scores ranging from 0 to 27. Higher scores indicate greater distress.
Patient Anxiety | Baseline, 7 weeks, 14 weeks, 26 weeks
  Patient anxiety will be measured using the Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 consists of 7 items, with total scores ranging from 0 to 21. Higher scores indicate greater anxiety.
Health-Related Quality of Life (St. George's Respiratory Questionnaire for COPD patients) | Baseline, 7 weeks, 14 weeks, 26 weeks
  Health-related quality of life will be measured using the St. George's Respiratory Questionnaire for COPD patients (SGRQ-C). The SGRQ-C consists of 40 items, with total scores ranging from 0 to 100. Higher scores indicate greater limitations and poorer health-related quality of life.
Health-Related Quality of Life (mMRC Dyspnoea Scale) | Baseline, 7 weeks, 14 weeks, 26 weeks
  Health-related quality of life will also be measured using the Modified Medical Research Council (mMRC) Dyspnoea Scale. The mMRC consists of 1 item, with a 5-point scale from 0 to 4. Higher scores indicate poorer health-related quality of life.
Health-Related Quality of Life (COPD Assessment Test™) | Baseline, 7 weeks, 14 weeks, 26 weeks
  Health-related quality of life will also be measured using the COPD Assessment Test™ (CAT™). The CAT consists of 8 items, with total scores ranging from 0 to 40. Higher scores indicate poorer health-related quality of life.
Time to COPD-Related Hospitalization | 12 months following enrollment
  Time to COPD-related hospitalization will be assessed by reviewing electronic health records for hospitalizations occurring within the 12-month period following enrollment. Hospitalizations will be identified as COPD-related if the condition is listed as a primary or secondary diagnosis, or if the records indicate that COPD was an active or contributory condition. Time to COPD hospitalization will be measured in days from the trial enrollment date.
All-Cause Mortality | 12 months following enrollment
  All-cause mortality will be tracked through electronic health record reviews. Additional data will be gathered from caregivers and confirmed through Internet obituary searches, if necessary, to ensure accurate capture of deaths not recorded in medical records.
Caregiver Burden | Baseline, 7 weeks, 14 weeks, 26 weeks
  Caregiver burden will be measured using the Zarit Caregiver Burden Inventory (ZBI). The ZBI consists of 22 items, with total scores ranging from 0 to 88. Higher scores indicate greater burden.
Family Relationship Quality | Baseline, 5 weeks, 12 weeks, 24 weeks
  Family relationship quality will be measured using the Family Emotional Involvement and Criticism Scale (FEICS). The FEICS consists of 14 items with 2 subscales (perceived criticism and emotional involvement), each with total scores ranging from 0 to 28. Higher scores indicate more expressed emotion in family relationships.
Self-Efficacy | Baseline, 5 weeks, 12 weeks, 24 weeks
  Self-efficacy will be measured among patients and caregivers using the General Self-Efficacy Scale (GSE). The GSE consists of 10 items, with total scores ranging from 10 to 40. Higher scores indicate greater self-efficacy.
Patient Loneliness | Baseline, 5 weeks, 12 weeks, and 24 weeks following enrollment
  Patient-reported loneliness will be measured using the UCLA Loneliness Scale. The UCLA Loneliness Scale consists of 20 items, with total scores ranging from 20 to 80. Lower scores indicate greater feelings of loneliness.
Caregivers' Psychological Distress | Baseline, 5 weeks, 12 weeks, 24 weeks
  Caregivers' psychological distress will be measured using the PHQ-9. As described above, the PHQ-9 consists of 9 items, with total scores ranging from 0 to 27. Higher scores indicate greater distress.
Caregiver Anxiety | Baseline, 5 weeks, 12 weeks, 24 weeks
  Caregivers' anxiety will be measured using the Generalized Anxiety Disorder-7 (GAD-7). As described above, the GAD-7 consists of 7 items, with total scores ranging from 0 to 21. Higher scores indicate greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Hart, MD, MSHP, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Henry Ford Health System, Detroit, Michigan
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Three datasets will be generated: (1) survey data from participants (patients and caregivers), (2) electronic health record data from patient participants, and (3) interview data from patients, caregivers, and clinicians. These datasets will be shared through the Inter-university Consortium for Political and Social Research (ICPSR) data repository. The shared data will be de-identified according to ICPSR's de-identification standards.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be made available as soon as possible or at the time of manuscript publication. The ICPSR allows for datasets to be archived and preserved on its servers indefinitely.
Access Criteria: Dataset A will be made available for public use via direct download from ICPSR, where usage will be free of charge to other ICPSR member institutions. Users who download the data are required to comply with ICPSR's Responsible Use Policy and must receive permission from ICPSR prior to re-distribution. Dependent on the stipulations of the data use agreements with HFHS, the investigators will enter into a restricted use agreement with ICPSR for resharing Dataset B under data use agreements and IRB permissions for the requestors. The investigators will be guided by ICPSR curators and the Penn IRB as to their assessment of the disclosure risk of Dataset C - even after deidentification of individual transcripts - to see if restricted use agreements are recommended.

DOCUMENTS (3):
  • Study Protocol (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT06600126/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT06600126/SAP_001.pdf
  • Informed Consent Form (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT06600126/ICF_002.pdf